CLINICAL TRIAL: NCT03185000
Title: A First in Human Feasibility Study of T Regulatory Cells (TR004) for Inflammatory Bowel Disease Using (ex Vivo) Treg Expansion
Brief Title: Treg Immunotherapy in Crohn's Disease
Acronym: TRIBUTE
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); Medical Research Council (Other Government); St. George's Hospital, London (Other); Miltenyi biotech (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRIBUTE Feasibility
Record Dates: First submitted 2017-04-13; First posted 2017-06-14 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — In Vitro Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immediate ATIMP (AP) (Experimental): Patients will receive Treg immunotherapy (TR004) infusion at Week 0.
  Interventions: Drug: TR004 (Treg immunotherapy)

INTERVENTIONS:
Drug: TR004 (Treg immunotherapy) — Administered Intravenously (IV)
  Other Names: Autologous regulatory T cells (Tregs) expanded in vitro

SUMMARY:
Crohn's Disease (CD) is a condition that causes inflammation of the digestive system or gut. Crohn's can affect any part of the gut, though the most common area affected is the end of the ileum (the last part of the small intestine), or the colon.

Crohn's is a chronic condition. This means that it is ongoing and life-long, although patients may have periods of good health (remission), as well as times when symptoms are more active (relapses or flare-ups).

Current available therapies frequently fail to maintain long-term remission and may be complicated by significant side effects.

There is an unmet medical need for novel therapies. Cellular therapies are emerging as potentially attractive therapeutic strategies.

The TRIBUTE trial will use autologous regulatory T cells (Tregs) expanded in vitro.

It is hoped that the administration of this treatment to patients with active CD will change the immune responses in the gut and reduce bowel wall inflammation.

DETAILED DESCRIPTION:
The TRIBUTE trial is looking at a new type of treatment for Crohn's Disease (CD), called regulatory T-cells (Tregs) immunotherapy.

Regulatory T-cells are naturally produced by the immune system. These cells have a powerful immunosuppressive action; they prevent auto-immune diseases by suppressing the over-active response that the immune system mounts against the body in these diseases. In addition it is thought that in patients with active CD, other immune cells in the gut are resistant to the normal controlling action of Tregs. Finally, we have found that Tregs that are isolated from patients and then are grown in the laboratory are more suppressive than Tregs freshly isolated from patients' blood.

Treg immunotherapy, TR004, will be unique to each patient. White blood cells will be extracted from their blood via leukapheresis. These cells will form the starting material to manufacture TR004 by expansion in a GMP accredited laboratory following a validated manufacturing process.

It will take approximately 23 days to produce enough cells for the immunotherapy treatment.

The trial aims to recruit a total of 4 patients diagnosed with moderate to severe CD. Men and women aged over 18 years who did not tolerate or did not respond to at least 2 standard treatments for the condition will be eligible to participate.

TRIBUTE is an open label first in human feasibility study of a single dose of TR004. Four participants will receive a single dose of TR004. Participants will be dosed singly. Safety data will be collected for five weeks post administration and reviewed by the DSMB before proceeding to dose the next participant. All participants will be followed up to week 21 to collect further safety and exploratory efficacy data, with additional safety monitoring at 1 and 2 years post dose. There is one dose level - 3.0 - 5.0 million TR004/kg.

Participants will be involved in the study for up to 24 months, from screening to safety follow-up at Week 104.

Eligible participants will receive one TR004 infusion at Week 0.

Patients will have a number of blood tests over the course of the trial. This will allow the doctors to monitor how safe TR004 is and how the body reacts to it.

Other tests, including vital signs such as blood pressure, heart rate and temperature, stool testing, and colonoscopy/biopsy will also be performed for this purpose and participants will have regular check-ups by the trial team. Scans such as CT scans, MRI scans or ultrasounds may be performed prior to starting the trial and participants will fill out questionnaires and diaries to monitor their progress over the course of the trial.

There are currently no known benefits to the participants in taking part in the study. While it is hoped that the treatment will reduce bowel inflammation, this may not happen. Participants may not directly benefit from taking part in this study but the information gained from their participation may help to improve the treatments available to other people with Crohn's Disease.

During the blood tests participants may experience discomfort and there is a risk of bleeding and bruising around the puncture site but this is very rarely serious.

During leukapheresis and on infusion day cannulas will be inserted in participant's veins. The cannula insertion may cause pain, bruising, or, on rare occasions, infection.

Some people find the leukapheresis uncomfortable due to having to stay in the same position for 2-3 hours. Blood calcium level may fall during the procedure and this can cause numbness and tingling in hands and feet and around the mouth. Patients can also feel cold, dizzy or sick.

A colonoscopy poses few risks. Rarely, complications of a colonoscopy may include:

* Reaction to the sedative used during the test
* Bleeding from the site where the tissue sample (biopsy) is taken
* A tear in the colon or rectum wall (perforation). The risk of this is less than 1 in 1,000.

This is the first time this particular expanded Tregs treatment will be tested in human so there may be potential unknown risks that could be serious. The anticipated risks of Treg administration are similar to those of a blood transfusion. The potential risks are likely to be lower because the cells infused will be the patient's own cells rather than cells from a blood donor. Common transfusion symptoms include a red, itchy skin rash, swelling of the hands, arms, feet, ankles and legs, dizziness and headaches. Less common symptoms include high temperature, chills and shivering.

The TRIBUTE study will be set-up and run at Guy's and St Thomas NHS Foundation Trust, London. It will be the only UK centre recruiting participants into the study.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent and able to comply with the protocol requirements
2. Male or female aged between 18 and 80 (inclusive) years of age at date of consent
3. A diagnosis of Crohn's disease (CD) established ≥12 weeks prior to date of consent by standard clinical, radiological, endoscopic and histological criteria
4. Documented moderate-to-severe CD with a Crohn's Disease Activity Index (CDAI) >= 220 within 3 months of date of consent
5. Active CD (mucosal inflammation) including ulceration, as assessed by colonoscopy at screening
6. Failure to tolerate or to respond to at least 2 prior lines of standard CD medication intended to induce or maintain remission, as determined by the referring gastroenterologist. Examples of such medications include, but are not limited to, azathioprine, mercaptopurine, methotrexate, vedolizumab, ustekinumab or anti-tumour necrosis factor antibody therapy. This does not include steroids and 5-ASA medications
7. Stable doses of concomitant medications
8. Normal or non-clinically significant electrocardiogram (ECG), as assessed by the Investigator at screening
9. Negative stool test for Clostridium difficile and faecal culture for standard pathogens at screening. For non-pathogenic organism, inclusion will be at the discretion of the Principal Investigator (PI)
10. Negative serology for HIV, Hepatitis B (cAb and sAg), Hepatitis C, HTLV and Syphilis at screening
11. Subject is judged by the principal investigator to be in otherwise good health based upon the results of all screening investigations in combination with medical history and physical examination

Exclusion Criteria:

1. A diagnosis of ulcerative colitis or IBD-unclassified
2. CD treatment-naïve patients, defined as patients who have never received or have refused standard CD treatment
3. History of clinically significant drug or alcohol abuse in the last 12 months prior to date of consent
4. Any history of major immune deficiency disorder, except Crohn's disease
5. Patients with a history of pulmonary embolism or deep vein thrombosis. Current or recent history (within 1 year prior to screening) of major organ or system failure or condition, acute or chronic that in the opinion of the investigator should preclude enrollment, except Crohn's disease
6. History of intestinal resection or intra-abdominal surgery within 6 months prior to date of consent
7. Requirement for immediate or imminent surgical, endoscopic or radiological intervention for indications including (but not limited to) toxic megacolon, obstruction, massive haemorrhage, perforation, sepsis, or intra-abdominal or perianal abscess
8. Patients with ileostomy or colostomy
9. Patients with short bowel syndrome (less than 1.5m of small bowel)
10. Complication of Crohn's disease such as strictures/stenosis, penetrating disease, or any other manifestation that might require surgery.
11. Patient has received therapeutic enema or suppository, other than required for endoscopy, within 14 days prior to date of consent and/or during the screening period
12. Patients who are currently using anticoagulants including but not limited to warfarin, heparin, enoxaparin, dabigatran, apixaban, rivaroxaban (note that anti-platelet agents such as aspirin up to 325mg daily or clopidogrel are permitted)
13. Use of corticosteroids on the day of leukapheresis sampling, prior to the procedure. Dosing should be delayed until after the procedure has been completed. This must be checked prior to the appointment and rescheduled if use is confirmed.
14. Current medically significant infection i.e. infection(s) requiring treatment with intravenous (IV) anti-infectives within 30 days prior to date of consent or oral anti-infectives for non-Crohn's disease related infections within 14 days prior to screening visit
15. Subject with an active systemic viral infection or any active viral infection that based on the investigator's clinical assessment makes the patient unsuitable for the study
16. History of tuberculosis (TB), unless there is documented evidence of completion of a full course of anti-TB treatment prior to screening. For patients with latent TB, as defined by a physician specialised in TB, they must have received prophylactic treatment for 4 weeks minimum prior to dosing
17. History of moderate to severe congestive heart failure (NYHA class III or IV), recent cerebrovascular accident (within 6 months of screening) and any other condition which, in the opinion of the investigator, would put the subject at risk by participation in the study
18. Subject with a previous history (within 12 months of consent) of dysplasia of the gastrointestinal tract, or found to have dysplasia in any biopsy performed during the screening endoscopy unless this is deemed to be a sporadic adenoma and has been completely removed
19. Significant laboratory abnormalities:

    Hb < 100g/L or WBC < 3.5 x 109/L or Plt < 100 x 109/L Creatinine > 1.5x ULN Total bilirubin > 34 µmol/L or ALT > 2x ULN or GGT > 2xULN. Elevated unconjugated bilirubin related to Gilbert's syndrome is allowed
20. Anti-TNF or ustekinumab therapy within 8 weeks of study dosing (day 0). Vedolizumab therapy within 5 half-lives (15 weeks) of dosing. Exposure to cyclosporine or tacrolimus within 2 weeks of date of consent
21. Patient currently receiving total parenteral nutrition (TPN) or plan to receive TPN at any time during the course of the study
22. Received another investigational drug within 60 days of anticipated study date of consent or 5 half lives whichever is greater
23. Patient who previously received stem cell transplantation
24. Current evidence of dysplasia or history of malignancy within the last 5 years of date of consent (except successfully treated squamous cell or basal cell carcinoma, without metastases or localised carcinoma in situ of the cervix)
25. Pregnant and lactating patients (females of childbearing potential with a positive serum pregnancy test at screening visit 1 or day -1 at week 0)
26. Female patients of childbearing potential (i.e. not post-menopausal or surgically sterilised) who are not willing to use effective methods of contraception (included but not limited to hormonal contraception, Intrauterine devices, sexual abstinence, vasectomised partner) to prevent pregnancy or abstain from heterosexual activity for the duration of the trial up to W21 visit
27. Male patients who are not willing to use an effective method of contraception (condoms) for the duration of the study up to W21 visit, when engaging in sexual activity with a female of childbearing potential
28. Allergy to any component / excipients used for the manufacture of TR004
29. Patient is considered by the investigator, for any reason, to be an unsuitable candidate for the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of dose-limiting toxicities (DLTs) | One period will be assessed, from Week 0 to Week 5
  Pre-defined safety events occurring within 5 weeks post-infusion

SECONDARY OUTCOMES:
Disease Activity Score (CDAI / PRO-2) calculated by evaluation of patient's diary completion and colonoscopy findings | CDAI / PRO-2 scores will be calculated at Week 0, Week 8, Week 21
  Measurement of clinical response
Biomarkers analysis (CRP, FCP) measured by blood test and stool sample analysis | CRP and FCP will be measured throughout the study, from Week 0 to Week 21
  Measurement of clinical response
Mucosal Healing Score (SES-CD) calculated by evaluation of colonoscopy findings | SES-CD scores will be calculated at screening and week 8
  Measurement of clinical response
Description of non-DLT adverse events | Week 0 to 5 and beyond week 5
  Pre-defined safety events occurring for the duration of the study

OTHER OUTCOMES:
Analysis of lymphocyte populations circulating in blood as well as localised in the intestinal lamina propria | Translational research samples will be collected at Week 1, 2, 3, 5, 9, 10, 11, 13, 16, 21
  Measurement of Immunological Response by analysis of translational research samples collected at specific time points.
  The baseline value will be compared to values obtained at subsequent time points, in order to measure the overall immunological response.
Cytokine levels in blood and in intestinal lamina propria | Translational research samples will be collected at Week 1, 2, 3, 5, 8,16, 21
  Measurement of Immunological Response by analysis of translational research samples collected at specific time points.
  The baseline value will be compared to values obtained at subsequent time points, in order to measure the overall immunological response.
Comparison of circulating and localised cells to determine differences and similarities | Translational research samples will be collected at Week 1, 2, 3, 5, 8,16, 21
  Measurement of Immunological Response by analysis of translational research samples collected at specific time points.
  The baseline value will be compared to values obtained at subsequent time points, in order to measure the overall immunological response.
Levels of circulating regulatory T cells labelled with Deuterium in blood | Translational research samples will be collected at Week 1, 2, 3, 5, 8,16, 21
  Measurement of Immunological Response by analysis of translational research samples collected at specific time points.
  The baseline value will be compared to values obtained at subsequent time points, in order to measure the overall immunological response.
Microbiome analysis from stool sample | Translational research samples will be collected at Week 1, 2, 3, 5, 8,16, 21
  Measurement of Immunological Response by analysis of translational research samples collected at specific time points.
  The baseline value will be compared to values obtained at subsequent time points, in order to measure the overall immunological response.
Feasibility - amount of TR0004 manufactured per patient | Between screening and dosing
  Dose level of TR004 therapy manufactured per patient
Feasibility - Number of participants recruited within the duration of the trial | Screening to Week 0 Day -1
  Number of participants that are enrolled into the study, confirmed as eligible at week 0 Day -1.
Feasibility - Number of study visits completed | From screening to week 104, including all study visits as defined in the protocol
  Number of study visits completed per patient recruited

CONTACTS AND LOCATIONS:
Overall Officials: Peter Irving, Dr, Principal Investigator — King's College London
Locations (1):
- Guy's Hospital - Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Canavan JB, Scotta C, Vossenkamper A, Goldberg R, Elder MJ, Shoval I, Marks E, Stolarczyk E, Lo JW, Powell N, Fazekasova H, Irving PM, Sanderson JD, Howard JK, Yagel S, Afzali B, MacDonald TT, Hernandez-Fuentes MP, Shpigel NY, Lombardi G, Lord GM. Developing in vitro expanded CD45RA+ regulatory T cells as an adoptive cell therapy for Crohn's disease. Gut. 2016 Apr;65(4):584-94. doi: 10.1136/gutjnl-2014-306919. Epub 2015 Feb 24. PMID 25715355
- [Derived] Rodger B, Clough J, Vasconcelos J, Canavan JB, Macallan D, Prevost AT, Lord GM, Irving P. Protocol for a first-in-human feasibility study of T regulatory cells (TR004) for inflammatory bowel disease using (ex vivo) Treg expansion (TRIBUTE). BMJ Open. 2025 Jan 23;15(1):e092733. doi: 10.1136/bmjopen-2024-092733. PMID 39855667
- [Derived] Goldberg R, Scotta C, Cooper D, Nissim-Eliraz E, Nir E, Tasker S, Irving PM, Sanderson J, Lavender P, Ibrahim F, Corcoran J, Prevost T, Shpigel NY, Marelli-Berg F, Lombardi G, Lord GM. Correction of Defective T-Regulatory Cells From Patients With Crohn's Disease by Ex Vivo Ligation of Retinoic Acid Receptor-alpha. Gastroenterology. 2019 May;156(6):1775-1787. doi: 10.1053/j.gastro.2019.01.025. Epub 2019 Jan 30. PMID 30710527
- See also: Related Info — http://gut.bmj.com/content/gutjnl/early/2015/02/24/gutjnl-2014-306919.full.pdf